CLINICAL TRIAL: NCT06726629
Title: Crosscultural Adaptation And Validation Of The Italian Version Of The New Knee Society Knee Scoring System
Acronym: KSS-ITALIAN
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: Ortopedia e Traumatologia - AO Ordine Mauriziano - Torino (Unknown); Traumatologia dello Sport - Campus Bio-medico- Roma (Unknown); Ortopedia e traumatologia - Policlinico di Modena (Unknown); Ortopedia e Traumatologia-Istituto IFCA Firenze (Unknown); Ortopedia e Traumatologia-Fondazione Poliambulanza Istituto Ospedaliero Brescia (Unknown)
Responsible Party: Sponsor
Other Study IDs: KSS-ITALIAN2023
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis
Keywords: KSS
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients
  Interventions: Other: Version Of The New Knee Society Knee Scoring System

INTERVENTIONS:
Other: Version Of The New Knee Society Knee Scoring System — All patients will be subjected to the same clinical and radiographic checks, the data of which will be collected in the different centres

SUMMARY:
The present study aims to be a multicenter prospective analysis aimed at validating the Italian version of the new KSS introduced in 2011 15. To do this it is first necessary to create the translation of the questionnaire. Several steps will be performed to obtain an adequate Italian version of the new KSS:

1. The English version of the KSS will be translated into Italian by 3 bilingual translators
2. The 2 versions will be submitted to the study collaborators (one per centre), the final version (accepted by all the study collaborators) will be translated back into English by 2 bilingual translators (native English) not aware of the initial version. The back translation will then be sent to the original author (Prof. Scott) to ensure that the consistency of the questionnaire has been maintained throughout all processes despite the necessary cultural adaptations.
3. Once the definitive version has been obtained, it will be tested by 300 Italian patients (with an estimated dropout of 20%) suffering from gonarthrosis. The patients will be distributed as follows: approximately 50 patients in each of the 6 centers (total 300). The number of patients was chosen considering approximately 17-18 patients for each of the 17 items, this choice is consistent with previously published studies on translation into other languages

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of gonarthrosis and indication for primary TKA surgery
* Age between 18 and 85 years
* Ability to respond to the proposed questionnaires and provide informed consent
* Availability for follow-up for one year after surgery

Exclusion Criteria:

* Concomitant hip or spinal problems, understood as a cause of patient discomfort even if not yet undergoing medical or rehabilitation therapy
* History of ipsilateral or contralateral knee surgery
* Congenital knee deformities
* Previous septic arthritis
* Neuromuscular pathology (e.g. polio)
* Simultaneous bilateral prosthesis or within 12 months of both knee, hip and ankle

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The analysis will be performed on all patients undergoing primary Total Knee Replacement (TKA) surgery at one of the centers included in the study
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
VALIDITY OF THE CONSTRUCT | at baseline (Day 0); post-operative (day 3), at 1 year follow-up
  Comparison between the Italian version of the KSS and the tests already validated in Italian .In particular, the Pearson or Spearman coefficient (depending on the sample distribution) will be used to evaluate the correlation.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Goh GS, Liow MHL, Bin Abd Razak HR, Tay DK, Lo NN, Yeo SJ. Patient-Reported Outcomes, Quality of Life, and Satisfaction Rates in Young Patients Aged 50 Years or Younger After Total Knee Arthroplasty. J Arthroplasty. 2017 Feb;32(2):419-425. doi: 10.1016/j.arth.2016.07.043. Epub 2016 Aug 10. PMID 27593732